CLINICAL TRIAL: NCT01758744
Title: TAPIT-1: Treatment of Pulmonary Hypertension Associated COPD With Inhaled Treprostinil-1
Brief Title: Treatment of Pulmonary Hypertension Associated COPD With Inhaled Treprostinil-1
Acronym: TAPIT-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-0560
Record Dates: First submitted 2012-12-06; First posted 2013-01-01 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Pulmonary Hypertension; COPD
Keywords: COPD PH; COPD associated Pulmonary Hypertension; COPD and Pulmonary Hypertension; Disease
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Disease, Chronic Obstructive; Disease | interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treprostinil (Experimental): Inhaled prostanoid therapy with Treprostinil
  Interventions: Drug: Inhaled Treprostinil Therapy

INTERVENTIONS:
Drug: Inhaled Treprostinil Therapy — Treprostinil: Inhaled prostanoid therapy
  Other Names: Tyvaso ®

SUMMARY:
An Open Label, Pilot Study Testing the Safety and Efficacy of Inhaled Treprostinil (Tyvaso®) in the Treatment of Pulmonary Hypertension (PH) Associated with Chronic Obstructive Pulmonary Disease (COPD)

DETAILED DESCRIPTION:
This is a pilot study of 10 patients that have COPD-PH. Primary outcome measure is to see if this drug is safe for this patient population and the secondary measure is to see if the drug improves patient functional capacity.

ELIGIBILITY:
Inclusion Criteria: must have:

* be between the ages of 30 and 80
* have a clinical diagnosis of Gold stage 2 to 4 COPD
* have a diagnosis of pulmonary hypertension established by a historic right heart catheterization
* a minimum weight of 45 Kg
* minimum systolic blood pressure of >90 mmHg
* be able to perform a six minute walk test
* be able to maintain a oxygen saturation >88% at rest (with or without oxygen)
* be treated with background therapy for COPD for a minimum of 1 month prior to consideration of enrollment.
* be competent to understand the information given in the Institutional Review Board (IRB) or Independent Ethics Committee (IEC) approved Informed Consent Form and must sign the form prior to the initiation of any study procedure.

Exclusion Criteria. Cannot have or be:

* The presence of pulmonary venous hypertension defined by a historical right heart catheterization
* Gold Stage I COPD
* documented left ventricular dysfunction as measured by echocardiography
* pregnant or breastfeeding
* Recipient of a lung transplant
* received chronic prostanoid therapy for pulmonary hypertension within 4 weeks prior to the screening appointment
* A requirement of greater than 9 l/min of O2 to maintain oxygen saturations greater than 88% at rest
* No other serious medical conditions

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
To assess the safety of Tyvaso ® as assessed by changes or stability of acute oxygenation (pulse oximetry) and spirometry (FEV1). | This is a 4 week trial
  A 4-Week, Open Label Study Testing the Safety of Inhaled Treprostinil (Tyvaso®) in the Treatment of Pulmonary Hypertension (PH) Associated with Chronic Obstructive Lung Disease (COPD) (PH-COPD)

SECONDARY OUTCOMES:
New York Heart Association (NYHA) functional class | Change in New York Heart Association (NYHA) functional class assessed at baseline and at week 4.
  A change in functional class is assessed as improvement or deterioration in the patient's functional status
Six minute walk distance | Change from baseline in 6 minute walk distance at 4 weeks
  A change in how far the subject can walk in 6 minutes will be measured at baseline and compared to how far the subject can walk in 6 minutes at week 4.
Clinical Worsening | From the time of randomization to until the subject discontinues from study for any cause, assessed up to 4 weeks
  Clinical worsening is described as Death, hospitalization (all cause)and COPD exacerbations (worsening of respiratory symptoms which require treatment with oral corticosteroids, antibiotics or both).
Peripheral Blood Mononuclear Cells (PBMC) phagocytic index (PI) and PBMC gene expression | Change from baseline in PBMC PI and PBMC gene expression at 4 weeks
  The phagocytic index is the average number of bacteria ingested per phagocyte in an incubated mixture of bacteria, phagocytes, and blood serum. We will also be looking a a change in gene expression of these (PBMC) cells.
  ------------------------------------------------------------------------------
St. George's Chronic Obstructive Pulmonary Disease (COPD) questionnaire | change from baseline in the St. George's respiratory questionnaire at 4 weeks
  The St. George's questionnaire is a quality of life questionnaire completed by the subject at baseline and at week 4.

CONTACTS AND LOCATIONS:
Overall Officials: Todd M. Bull, M.D., Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Denver, Aurora, Colorado
  - University of Florida College of Medicine, Jacksonville, Florida